CLINICAL TRIAL: NCT01251159
Title: Somatic Mutations in Stem and Progenitor Cells in AML
Brief Title: Biomarkers in Bone Marrow Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000688223; ECOG-E1900T4
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Polymerase Chain Reaction; Immunologic Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: immunologic technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is studying bone marrow samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To rigorously examine fractionated hematopoietic stem and progenitor cells from patients with acute myeloid leukemia (AML).
* To define somatic mutations occurring in de novo AML, including the FLT3-ITD, CEBPA, NPM1, TET2, ASXL1, IDH1, and IDH2 mutations.
* To examine what cellular compartments (LT-HSC, ST-HSC, CMP, GMP, and MEP) contain the selected mutations and in what order those mutations occur.

OUTLINE: Archived bone marrow specimens are analyzed for sequencing and detection of mutations by Sanger-based resequencing of PCR amplicons. Results are then compared with the results of age-matched healthy controls.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Bone marrow samples must meet 1 of the following criteria:

  * Normal karyotype from patients enrolled on ECOG-1900 archived at the ECOG Leukemia Tissue Bank

    * Live, sortable mononuclear cells prepared at the time of initial diagnosis (slow-frozen in media with 10% DMSO OR fresh cells shipped immediately
  * Age-matched healthy control samples from commercial providers

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Samples from patients enrolled on E1900 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-05-15 (Actual); Primary Completion 2009-06-15 (Actual); Study Completion 2009-06-15 (Actual)

PRIMARY OUTCOMES:
Define somatic mutations occurring in de novo AML | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich G. Steidl, MD, BS, Principal Investigator — Albert Einstein College of Medicine